CLINICAL TRIAL: NCT00045123
Title: Phase IIB, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Efficacy of MPC-7869 in Delaying the Systemic Progression of Prostate Cancer in Patients With Intermediate to High Risk of Recurrence With Rising PSA Levels After Prostatectomy, Prostatectomy and Radiotherapy or Radiotherapy Alone for Localized Disease
Brief Title: R-Flurbiprofen in Treating Patients With Localized Prostate Cancer at Risk of Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Myrexis Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000256371; MYRIAD-MPR-7869-001; NCT00043251 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-02-06 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tarenflurbil; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: tarenflurbil
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. R-flurbiprofen may be effective in delaying the recurrence of localized prostate cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of R-flurbiprofen in treating patients who have localized prostate cancer at risk of recurrence following radiation therapy and/or prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of R-flurbiprofen on time to systemic disease progression evaluated over a minimum of 3 years in patients with localized adenocarcinoma of the prostate with an intermediate or high risk of recurrence and rising prostate-specific antigen (PSA) levels after radiotherapy alone, prostatectomy alone, or both radiotherapy and prostatectomy.
* Determine the effect of this drug on the change in serum PSA levels over time prior to androgen-deprivation therapy (ADT) in these patients.
* Determine the effect of this drug on the time of initiation of ADT in these patients.
* Determine the effect of this drug on the number of patients requiring ADT.
* Determine the safety of this drug in these patients.
* Determine the population pharmacokinetics of R-flurbiprofen and bioinversion of R-ToS in this patient population.
* Determine the number of patients with systemic disease progression at the end of the study.
* Determine the time to clinical disease progression in patients treated with this drug.
* Determine the time to prostate cancer-related mortality and time to all cause mortality in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to risk of recurrence based on Gleason score at diagnosis (5-7 vs 8-10). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral low-dose R-flurbiprofen twice daily.
* Arm II: Patients receive oral high-dose R-flurbiprofen twice daily.
* Arm III: Patients receive oral placebo twice daily. In all arms, treatment continues for up to 5.5 years (66 months) in the absence of disease progression or unacceptable toxicity. Patients who demonstrate increased prostate-specific antigen without objective disease progression and require androgen-deprivation therapy (ADT) continue receiving R-flurbiprofen. Patients who develop local recurrence or systemic disease may withdraw from study and receive additional therapy off study.

PROJECTED ACCRUAL: Approximately 390 patients (130 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed localized adenocarcinoma of the prostate (from a pre-operative core biopsy, surgical specimen, or post-therapy core biopsy)
* Gleason score 5-10 at diagnosis (the highest score is used if multiple scores are available)
* Must have undergone 1 of the following curative treatment strategies:

  * Radical prostatectomy

    * Not a candidate for radiotherapy
  * Radical prostatectomy followed by radiotherapy at the time of surgery or any time thereafter
  * Radiotherapy of the prostate and/or surrounding structures by external beam radiotherapy (EBRT), brachytherapy (BT), or a combination of EBRT and BT
* Must have 3 consecutive rising prostate-specific antigen (PSA) measurements OR meets slope criteria
* Biochemical failure, meeting 1 of the following criteria:

  * PSA at least 0.2 ng/mL post radical prostatectomy
  * PSA greater than 1.5 ng/mL after radiotherapy or appropriate calculated slope
* Testosterone at least 100 ng/mL
* No rise in PSA with concurrent clinically active prostatitis
* No metastatic prostate cancer
* PSA no greater than 20.0 ng/mL

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST or ALT no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No uncontrolled cardiac conditions
* No New York Heart Association class III or IV heart disease

Gastrointestinal

* No active ulcer disease diagnosed within the past 3 months
* No upper gastrointestinal bleed requiring a transfusion within the past 3 years
* No non-steroidal anti-inflammatory drug (NSAID)-associated ulcers within the past 5 years

Other

* No known hypersensitivity to NSAIDs, including COX-2-specific inhibitors (e.g., celecoxib or rofecoxib)
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer
* No active systemic infections
* No other serious uncontrolled medical condition
* No dementia or altered mental status

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* More than 5 years since prior cytotoxic chemotherapy for other malignant disease
* No prior cytotoxic chemotherapy for prostate cancer
* No concurrent chemotherapy

Endocrine therapy

* More than 9 months since prior androgen-deprivation therapy other than as cytoreductive therapy (neoadjuvantly or adjuvantly for less than 9 months) with the intent to cure
* More than 3 months since prior cyproterone, finasteride, diethylstilbestrol, megestrol, or other hormonally active (antiandrogen or antiprostate) therapies

Radiotherapy

* See Disease Characteristics
* No prior strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium, or other radioisotope materials for palliative intent or metastasis intervention
* Concurrent iodine I 125 or palladium Pd 103 for primary brachytherapy with curative intent allowed

Surgery

* See Disease Characteristics
* More than 8 weeks since prior major surgery and recovered
* No prior orchiectomy

Other

* More than 1 month since prior PC-SPES
* More than 1 month since prior investigational agents or devices (6 months for other investigational therapy for prostate cancer)
* No prior bisphosphonates (e.g., pamidronate, alendronate, or clodronate) for palliative intent or metastasis intervention
* At least 2 months since prior chronic non-steroidal anti-inflammatory drugs (NSAIDs), including cyclooxygenase-2 (COX-2)-specific inhibitors (e.g., celecoxib or rofecoxib), administered for more than 7 days per month
* No concurrent CYP2C9 inhibitor or substrates, including but not limited to the following:

  * Phenytoin
  * Fluvastatin
  * Amiodarone
  * Fluconazole
  * Acenocoumarol
  * Diclofenac
* No concurrent ketoconazole
* No concurrent antiretroviral therapy for HIV-positive patients
* Concurrent cardioprotective aspirin up to 100 mg once daily allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Sheron B. Bass, RN, MS — Myrexis Inc.
Locations (58):
- United States (58):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Urology Associates Of Central California, Fresno, California
  - Orange County Urology Associates, Laguna Hills, California
  - South Orange County Hematology-Oncology Associates, Laguna Hills, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Atlantic Urology Medical Group, Long Beach, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - San Diego Urological Medical Group, San Diego, California
  - Coastal Medical Research Group, Incorporated, San Luis Obispo, California
  - Urology Associates - Research, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - UroSearch - Ocala, Ocala, Florida
  - Rice, Lake and Harper Urology, LLC, Columbus, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Cancer Care Specialists of Central Illinois, S.C. - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Regional Urology, L.L.C., Shreveport, Louisiana
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Drs. Werner, Murdock and Francis, P.A., Urology Associates, Greenbelt, Maryland
  - Lakeside Urology, P.C., Saint Joseph, Michigan
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Las Vegas, Nevada
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Center for Urologic Care, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - AccuMed Research Associates, Garden City, New York
  - Staten Island Urologic Oncology, Staten Island, New York
  - Urology Center, Greensboro, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Urological Associates, Incorporated, Columbus, Ohio
  - Oregon Urology Specialists, Eugene, Oregon
  - Center for Urologic Care, Bryn Mawr, Pennsylvania
  - Urological Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Center of Urologic Care of Berks County, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University Urological Research Institute, Providence, Rhode Island
  - Grand Strand Urology LLP, Myrtle Beach, South Carolina
  - University of Tennessee - Graduate School of Medicine, Knoxville, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Urology Consultants, P.A., San Antonio, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Northwest Hospital and Medical Center, Seattle, Washington
  - Highline Hospital Campus, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin